CLINICAL TRIAL: NCT02500602
Title: CAP - Doxazosin in the Treatment of Co-Occurring PTSD and Alcohol Use Disorders
Brief Title: CAP: Doxazosin in the Treatment of Co-Occurring PTSD and Alcohol Use Disorders
Acronym: Doxazosin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLE-001-14F; CX001288 (Other Grant/Funding Number: VA/DoD); NCT02492334 (obsolete NCT alias)
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Posttraumatic Stress Disorder; Alcohol Use Disorders
Keywords: PTSD; alcohol use disorders; posttraumatic stress disorder; AUD; Veteran; substance use disorders; SUD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxazosin (Experimental): Participants randomly assigned to receive doxazosin (target dose of 16 mg/day). Doxazosin will be initiated at 1 mg/day for the first week, 2mg/day for the second week, 4mg/day for the third week, 8mg/day for the fourth week, and then increase to 16 mg/day for the remaining eight weeks (as tolerated). Research staff administered the study medication at the weekly visits, and participants were given take-home doses of the medication to self-administer on the days in between study visits.
  Interventions: Drug: doxazosin
- Placebo (Placebo Comparator): Participants randomly assigned to placebo. Research staff administered the study medication at the weekly visits, and participants were given take-home doses of the medication to self-administer on the days in between study visits.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: doxazosin — active medication
  Arms: Doxazosin
Drug: placebo — placebo pill
  Arms: Placebo

SUMMARY:
The proposed study will examine the efficacy of doxazosin in the treatment of PTSD and alcohol use disorder or substance use disorders.

DETAILED DESCRIPTION:
Due to sustained military conflicts in Afghanistan and Iraq over the past decade, there are an increasing number of U.S. military personnel and Veterans returning home with posttraumatic stress disorder (PTSD) and comorbid alcohol use disorders (AUD) and substance use disorders (SUD). If left untreated, Veterans with co-occurring PTSD and substance use disorders are at increased risk for developing other mental health problems (e.g., depression, anxiety), suicidal ideation and attempts, physical health problems, reduced resiliency and military readiness, employment problems, violence, and family/relationship impairment. While mental health services are in place for U.S. service members, substantial gaps in the treatment of co-occurring PTSD and SUD exist and there is little scientific evidence available to guide the provision of care. As part of the Consortium to Alleviate PTSD (CAP), the proposed study directly addresses this critical knowledge gap by testing the efficacy of doxazosin, a long-acting and selective alpha-1 adrenergic antagonist, as compared to placebo in reducing PTSD and AUD/SUD severity among U.S. military personnel. The medication to be investigated (doxazosin) represents a novel treatment approach for PTSD and AUD/SUD. While prazosin, also an alpha-1 adrenergic antagonist, has been shown to improve sleep and nightmares in military personnel with PTSD and may help reduce substance use severity, it has a short half-life of 2-3 hours and requires multiple doses each day, which is a significant limitation. In several pilot studies, doxazosin has shown promise in significantly reducing symptoms of PTSD and AUD/SUD and, in contrast to prazosin, it requires once per day dosing which confers a significant advantage in terms of translating positive findings into routine clinical practice. In this Stage II study, the investigators will (1) employ a two-arm randomized, double-blind, between-groups experimental design that will consist of 12 weeks of treatment with doxazosin or placebo medication; (2) use standardized, repeated dependent measures to rigorously assess PTSD symptomatology and AUD/SUD severity; (3) measure impairment in associated mental and behavioral health problems (e.g., depression, anxiety, sleep, risky behaviors, family/social functioning); and (4) use functional magnetic resonance imaging (fMRI) to investigate the underlying pathophysiology of comorbid PTSD/AUD and identify prognostic indicators of treatment outcome. To achieve these aims, the investigators have assembled a multidisciplinary team of investigators with nationally-recognized expertise in combat-related PTSD, substance use disorders and neuroimaging who have successfully collaborated in the past and are uniquely qualified to implement this type of investigation. The investigators represent a collaboration of faculty at the Ralph H. Johnson Veterans Affairs (VA) Medical Center and the Medical University of South Carolina (MUSC) in Charleston, SC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; any race or ethnicity.
2. Served in U.S. Military - any branch or operation.
3. Subjects must be able to comprehend English.
4. Meet criteria for current (i.e., last 6 months) Substance Use Disorder (SUD) using a modified version of the MINI 7.0 (i.e., must meet DSM-5 criteria for SUD in the past 6 months instead of 12 months).
5. Meet DSM-5 criteria for current (i.e., last month) PTSD.
6. Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before treatment initiation. This is because initiation or change of medications during the course of the trial may interfere with interpretation of results.
7. Must consent to random assignment to doxazosin or placebo.
8. Must consent to complete all treatment and follow-up visits.

Exclusion Criteria:

1. Subjects meeting DSM-5 criteria for current bipolar affective disorders, as the study protocol may be therapeutically insufficient.
2. Subjects experiencing significant withdrawal symptoms, as evidence by a score of 10 or above on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA). These subject will be referred for clinical detoxification and may be re-assessed for study eligibility after medically supervised detoxification has been completed.
3. Individuals considered an immediate suicide risk or who are likely to require hospitalization during the course of the study.
4. Previous treatment with doxazosin.
5. Subjects on maintenance anxiolytic, antidepressant, or mood stabilizing medications which have been initiated during the past four weeks. If it is determined, based on clinical criteria, that a subject needs to be started on maintenance medications for anxiety, mood or psychotic symptoms during the course of the study, they may be discontinued from the treatment trial.
6. Women who are pregnant, nursing or not practicing an effective form of birth control.
7. Individuals with a history of or current medical illness including unstable angina, myocardial infarction, congestive heart failure or other cardiac condition, hypotension, renal or hepatic disorders, endocrine disorders, prostate or other cancer, pancreatitis, or a seizure disorder.
8. Subjects with abnormal liver function test (LFTs) as evidenced by laboratory findings of SGOT or SGPT greater than two times normal.
9. Subjects with a history of adverse reactions to quinazolines or other alpha-1-antagonists (such as allergic reactions, priapism, hepatitis, angioedema, or intraoperative floppy iris syndrome).
10. Individuals currently taking alpha blockers (terazosin, prazosin), hypnotics/benzodiazepines, atypical antipsychotics (olanzapine, quetiapine, risperidone, clozapine), alpha-2-agonists (Clonidine, methyldopa, tizanidine, guanfacine), conivaptan, boceprevir, idelalisib, PDE-5 inhibitors or alpha-1-antagonists, protease inhibitors (treatment of HIV), oral antifungals, alfuzosin, pazopanib, silodosin, tadalafil, or tamulosin.
11. MRI exclusions: Claustrophobia; tattoos above the shoulders after evaluation by MRI technician; permanent eyeliner or permanent artificial eyebrows; cardiac pacemaker; metal fragments in eye, skin, or body, including shrapnel; heart valve replacement; brain clips; venous umbrella; being a sheet-metal worker or welder; lifetime history of aneurysm surgery; intracranial bypass, renal, or aortic clips; prosthetic devices such as middle ear, eye, joint, or penile implants; joint replacements; non-removable hearing aid, neurostimulator, or insulin pump; shunts/stents; metal mesh/coil implants; metal plate/pin/screws/wires; or any other metal implants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudie E. Back, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Plan: The data collected from study participants, including PHI, will be entered into and securely stored in the STRONG STAR-CAP database on a secure UTHSCSA server by a member of the study research team under a signed Data Use Agreement between Ralph H. Johnson VA and UTHSCSA. Terms of the Data Use Agreement data have been reviewed and approved by VACO and found to meet VA security compliance standards. Electronic data will be stored, managed, and analyzed by the Data Management and Biostatistics Core staff of the STRONG STAR-CAP Consortium. The overall study PI and named collaborators will have access to identifiable data through the STRONG STAR-CAP website and UTHSCSA server.
Supporting Information: ICF

REFERENCES:
- [Derived] Back SE, Flanagan JC, Mintz J, Brady KT, Jones J, Jarnecke AM, Joseph JE, Shirley DW, Malcolm RJ, Hamner M, Litz BT, Niles BL, Young-McCaughan S, Keane TM, Peterson AL. A Double-Blind Randomized Controlled Trial of Doxazosin for Co-Occurring PTSD and Alcohol Use Disorder in Veterans. J Clin Psychiatry. 2023 Mar 8;84(2):21m14367. doi: 10.4088/JCP.21m14367. PMID 36883885

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxazosin: Participants randomly assigned to receive doxazosin (target dose of 16 mg/day).
  doxazosin: active medication
- Placebo: Participants randomly assigned to receive Placebo pill
  placebo: placebo pill
Period: Treatment Phase
Arm/Group | Doxazosin | Placebo
Started | 74 | 70
Completed | 68 | 69
Not Completed | 6 | 1
Period: Follow Up Phase
Arm/Group | Doxazosin | Placebo
Started | 68 | 69
Completed | 53 | 47
Not Completed | 15 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxazosin | Placebo | Total
Number analyzed (Participants) | 74 | 70 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.9) | 45.5 (11.4) | 45.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 60 | 62 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 34 | 36 | 70
  White | 33 | 29 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 70 | 144

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale
Description: The primary PTSD outcome measure was the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013). The CAPS-5 is a semi-structured interview that measures the DSM-5 symptoms of PTSD and requires the presence of at least one intrusion symptom, one avoidance symptom, two cognition and mood symptoms, and two arousal symptoms for a period of 1 month or more to reach diagnostic threshold. There are 20 symptom items and responses that are rated on a 5-point scale ranging from 0 (absent) to 4 (extreme/incapacitating), with a total PTSD symptom severity score of the sum of the 20 symptom items ranging from 0-80, and lower scores indicating better outcomes (or less severe PTSD symptomology). The CAPS-5 was assessed at end of treatment (week 12).
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Doxazosin: Doxazosin (target dose of 16 mg/day). Doxazosin will be initiated at 1 mg/day for the first week, 2mg/day for the second week, 4mg/day for the third week, 8mg/day for the fourth week, and then increase to 16 mg/day for the remaining eight weeks (as tolerated). R
  doxazosin: active medication
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 74 | 70
score on a scale | 34.2 (9.6) | 32.5 (8.7)

2. Primary Outcome: PTSD Checklist (PCL-5)
Description: The secondary PTSD outcome measure was the PTSD Checklist-5 (PCL-5; Weathers et al., 2013b). The PCL-5 is 20-item self-report measure that assesses the DSM-5 symptoms of PTSD using a severity rating Likert scale ranging from 0 to 4 that indicates the degree of distress across symptoms (0 = not at all to 4 = extremely). The overall score range is 0-80 (and combines the score for all 20 symptoms), with lower scores representing better outcomes (less severe PTSD symptomology). The PCL-5 was assessed at end of treatment (week 12).
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 74 | 70
score on a scale | 47.3 (14.5) | 46.9 (15.2)

3. Primary Outcome: Time Line Follow Back (TLFB)
Description: The TLFB obtains retrospective self-report of substance use by using a calendar and memory prompts to stimulate recall (Sobell & Sobell, 1992). Quantity and frequency assessments are made using this instrument (e.g., total number of standard drink units, percent of days using) as well as abstinence (yes/no). TLFB yields consistently high test-retest correlations and correlates well with other self-reports and collateral reports (Sobell et al., 2003). The TLFB assesses frequency and amount of substance use over a pre-determined timeframe. TLFB data were collected throughout the trial, and the values reported here represent the TLFB data at end of treatment (week 12).
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 74 | 70
percent
  percentage of days drinking | 53.7 (34.8) | 48.1 (41.2)
  percent heavy days drinking | 37 (37.6) | 38.6 (38)

ADVERSE EVENTS:
Time Frame: AEs collected from baseline (if baseline lasted longer than one appointment) through follow up (12 week treatment phase and 6 week follow up - approximately 20 weeks)
Description: Participants were asked about any changes in health or existing symptoms at each visit.
Arm/Group | Doxazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/70
Serious Adverse Events (participants affected / at risk) | 12/74 | 9/70
Other Adverse Events (participants affected / at risk) | 48/74 | 40/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxazosin (N=74) | Placebo (N=70)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — Pt experienced chest pain and was sent to ER by PCP, admitted to hospital for 2 days. Event occurred prior to any medication administration.
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) — Internal hemorrhoids
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Pancreatitis
Dehydration (General disorders) | 1 (1) | 0 (0) — Participant admitted to hospital for dehydration secondary to viral gastroenteritis
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant fell while running, fractured left shoulder
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation/Attempt (Psychiatric disorders) | 3 (3) | 1 (1)
Anger/Frustration (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal Ideation/Aggression (Psychiatric disorders) | 1 (1) | 1 (1) — Placebo - participant reported feeling extreme anger related to housing. Reported 'intent to harm others' to police in order to be admitted to hospital. Dox-Participant expressed homicidal ideation towards VA security guard and MD
Substance Use (Psychiatric disorders) | 1 (1) | 3 (3)
Panic Attack/Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetes Complications (Endocrine disorders) | 1 (1) | 1 (1) — Dox - Diabetes mellitus with metabolic acidosis Placebo - insulin stopped working
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxazosin (N=74) | Placebo (N=70)
Depression (Psychiatric disorders) | 7 (7) | 5 (5)
Hypotension (Cardiac disorders) | 0 (0) | 4 (4)
Hypertension (Cardiac disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Stomach Virus/Cramping/Nausea (Gastrointestinal disorders) | 13 (13) | 6 (6)
Cold/Sinus/Congestion (General disorders) | 7 (7) | 14 (14)
Fatigue (General disorders) | 2 (2) | 5 (5)
Generalized Pain (General disorders) | 5 (5) | 3 (3)
Accident/Injury (General disorders) | 8 (8) | 4 (4)
Joint/Muscle Pain (Metabolism and nutrition disorders) | 11 (11) | 16 (16)
Drowsiness/Grogginess (Nervous system disorders) | 11 (11) | 6 (6)
Dizziness/Lightheadedness (Nervous system disorders) | 9 (9) | 19 (19)
Sleep Problems (Psychiatric disorders) | 10 (10) | 10 (10)
Vivid Dreams/Nightmares (Psychiatric disorders) | 8 (8) | 12 (12)
Emotional Distress (Psychiatric disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02500602/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT02500602/ICF_000.pdf